CLINICAL TRIAL: NCT04497896
Title: Epidemiology, Aetiologies, and Complications of Playtime Open-globe Injuries in Children
Brief Title: Playtime Open Globe Injuries in Children
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300438
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Eye Trauma
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Repair of open globe injury — repair of corneal, corneoscleral, or scleral wounds

SUMMARY:
This study investigated the epidemiology, aetiologies, and complications of playtime open-globe injuries in children at the Assiut University Hospital, Egypt, between January to July 2016.

DETAILED DESCRIPTION:
This prospective study was conducted at the Department of Ophthalmology, Assiut University Hospital, which is the largest tertiary referral hospital in Upper Egypt and provides 24-hour ophthalmic emergency services for six governorates. The study included all children (age ≤18 years) admitted with open-globe injuries that occurred during playtime over a 6-month study period. Demographic information (age and sex), the site and mechanism of injury, the site of ocular laceration (corneal, scleral or corneoscleral) and associated complications were recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* all children (age ≤18 years) admitted with open-globe injuries that occurred during playtime over a 6-month study period (January-July 2016).

Exclusion Criteria:

* Open globe injuries in patients olader than 18 years.
* Closed globe injuries

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: all children (age ≤18 years) admitted to Assiut university hospital with open-globe injuries that occurred during playtime over a 6-month study period (January-July 2016).
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity (in Decimal using Snellen chart) after repair of open globe injury | 1 day
  measurement of corrected distant visual acuity after wound repair.

IPD SHARING:
Plan to Share IPD: No